CLINICAL TRIAL: NCT03995927
Title: Palliative Radiation Oncology Chief's Clinic (PROCC): Assessing the Impact of a Dedicated Clinic on the Timeliness of Palliative Radiotherapy
Brief Title: Palliative Radiation Oncology Chief's Clinic
Acronym: PROCC
Status: Terminated | Type: Observational
Why Stopped: PI decision, technical events unrelated to study slowing down the process and ability to accrue
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00058996; WFBCCC 03419 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Malignant Disease; Metastasis
Keywords: Difficult to treat cancers
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data collection/questionnaire: Data collection for patient medical charts and patient fill out questionnaires first visit and post-treatment visits
  Interventions: Other: Data collection and analysis; Other: Quality of Life Questionnaire

INTERVENTIONS:
Other: Data collection and analysis — Only radiation oncology patients data from medical records regarding treatment, demographics and follow-up visits will be collected and logged by investigators.
Other: Quality of Life Questionnaire — Participants will be asked to complete a set of short forms at first visit and post-treatment visits. If participant has a routine visit about 3 months after treatment, participant will be asked to complete a final form that is optional.

SUMMARY:
The proposed study represents a quality improvement study of a recently-developed dedicated radiation oncology subspecialty clinic with the goal of improving timeliness of palliative radiation therapy and improving resident training in palliative care topics. The aim of this study is to evaluate the impact of this clinic on time to palliative radiation therapy following referral.

DETAILED DESCRIPTION:
Primary Objective:

• Determine whether interval between palliative radiation therapy referral and palliative radiation therapy initiation is shorter for participants treated in a dedicated palliative radiation oncology clinic compared to the same interval for participants treated in a general radiation oncology clinic (historical control). The investigators' hypothesis is that this interval will be significantly shorter among the Palliative Radiation Oncology Chief's Clinic participants compared to historical control.

Secondary Objectives:

* Determine whether each of the three component intervals within the overall interval from referral to treatment initiation (i.e., referral to consultation; consultation to simulation; simulation to treatment) is shorter for participants treated in a dedicated palliative radiation oncology clinic compared to the length of the same intervals for participants treated in a general radiation oncology clinic (historical control). The investigators' hypothesis is that each of these component intervals will be significantly shorter among the Palliative Radiation Oncology Chief's Clinic participants compared to historical control.
* Describe levels of and changes over time in patient-reported quality of life after palliative radiation therapy in the full sample, and in subgroups stratified by various radiation regimens. The investigators' hypothesis is that participants who receive a shorter course of palliative radiation (one day or five days) will have greater improvements in overall quality of life than participants who receive a ten-day course of palliative radiation.
* Determine median overall survival after palliative radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinically or pathologically-defined malignant disease amenable to palliative radiotherapy.

Exclusion Criteria:

* Pregnancy. A verbal pregnancy denial will suffice.
* No intention to treat with palliative radiation therapy following initial referral and consult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of patients referred to radiation oncology for consideration of palliative radiation therapy
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Number of Days Between Referral and Start of Treatment | 3 months
  Number of days between referral to palliative radiation therapy interval and start of palliative radiation therapy compared to historical control. Mean time from referral to the start of RT (measured in days) will be computed for our sample and compared to the historical control mean of 13.4 days using a two-sided one-sample t-test.

SECONDARY OUTCOMES:
Mean Time from Referral for Consultation | 3 months
  Mean time from referral to consultation will be computed for our sample and compared to the historical control mean of 3.6 days.
Mean Time from Consultation to CT Simulation | 3 months
  Mean time from consultation to CT simulation will be computed for our sample and compared to the historical control mean of 3.8 days.
Mean Time from CT Simulation to Palliative Radiation Start | 3 months
  Mean time from CT simulation to start of PRT will be computed for our sample and compared to the historical control mean of 6.1 days.
Quality of Life Changes | 1 and 3 months after treatment completion
  Levels of and changes in patient-reported overall quality of life as measured by the EORTC QLQ-C15-PAL (14 questions) at baseline and at 1-month and 3-month intervals after end of palliative radiation therapy. Quality of life score scale consists of 1 = not at all to 4 = very much. The higher the QOL score the greater change in the participant's quality of life.
Overall Survival | 6 months after treatment completion
  Median overall survival (number of days between start of radiation therapy and death from any cause) will be estimated using the Kaplan-Meier method and compared (with a one-sample logrank test and assuming a Weibull distribution parameter of 1.0) to the median overall survival of n=134 days in our historical control.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Brown, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No